CLINICAL TRIAL: NCT01655628
Title: Autologous Cytokine-Induced Killer Cell Transfusion in Combination With Gemcitabine Plus Cisplatin Regimen Chemotherapy for Metastatic Nasopharyngeal Carcinoma
Brief Title: GC Regimen Chemotherapy Plus CIK Cells for Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian-jun Li, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120704
Record Dates: First submitted 2012-07-26; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Stage IV Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; metastasis; gemcitabine; CIK cells
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GC chemotherapy plus CIK cells (Experimental): A total of 40 patients enrolled will be accept 4 cycles GC chemotherapy(every 4 weeks),then they will randomized divided into two groups. 20 patients will maintain autologous CIK cells for 8 cycles (every 4 weeks); however,the other 20 patients will not accept CIK cells treatment. After the all 40 patients have accomplished 4 cycles GC regimen chemotherapy plus 8 cycles CIK cells treatment or 4 cycles GC chemotherapy alone, the early effects will be assessed and long-term efficacy such as OS and PFS will be evaluated.
  Interventions: Drug: GC chemotherapy plus CIK cells (Gemcitabine, Cisplatin, Autologous CIK cells)
- GC chemotherapy (Active Comparator): A total of 40 patients enrolled will be accept 4 cycles GC chemotherapy(every 4 weeks),then they will randomized divided into two groups. 20 patients will maintain autologous CIK cells for 8 cycles (every 4 weeks);the other 20 patients will not accept CIK cells treatment. After the all 40 patients have accomplished 4 cycles GC regimen chemotherapy plus CIK cells treatment or 4 cycles GC chemotherapy alone, the early effects will be assessed and long-term efficacy such as OS and PFS will be evaluated.
  Interventions: Drug: GC chemotherapy (Gemcitabine, Cisplatin)

INTERVENTIONS:
Drug: GC chemotherapy plus CIK cells (Gemcitabine, Cisplatin, Autologous CIK cells) — A total of 40 patients enrolled will be accept 4 cycles GC chemotherapy(every 4 weeks),then they will randomized divided into two groups. 20 patients will maintain autologous CIK cells for 8 cycles (every 4 weeks);the other 20 patients will not accept CIK cells treatment. Afer the all 40 patients have accomplished 4 cycles GC regimen chemotherapy plus CIK cells treatment or 4 cycles GC chemotherapy alone, the early effects will be assessed and long-term efficacy such as OS and PFS will be evaluated.
  Other Names: Gemcitabine (Zefei) and Cisplatin(Nuoxin) ;; Autologous CIK cells
  Arms: GC chemotherapy plus CIK cells
Drug: GC chemotherapy (Gemcitabine, Cisplatin) — A total of 40 patients enrolled will be accept 4 cycles GC chemotherapy(every 4 weeks),then they will randomized divided into two groups. 20 patients will maintain autologous CIK cells for 8 cycles (every 4 weeks);the other 20 patients will not accept CIK cells treatment. Afer the all 40 patients have accomplished 4 cycles GC regimen chemotherapy plus CIK cells treatment or 4 cycles GC chemotherapy alone, the early effects will be assessed and long-term efficacy such as OS and PFS will be evaluated.
  Other Names: Gemcitabine (Zefei) and Cisplatin (Nuoxin)
  Arms: GC chemotherapy

SUMMARY:
Nasopharyngeal carcinoma (NPC) is one of the most common malignant tumors in Southern China and South Asia. After radiotherapy, some patients with nasopharyngeal carcinoma still had distant metastasis. In recent years, some chemotherapeutic agents, such as gemcitabine, cisplatin, were used to treat patients with advanced nasopharyngeal carcinoma, including those with local recurrence and distant metastases, with a certain short-term effect. However, chemotherapy alone is still not ideal for effectively improving the prognosis of patients with advanced nasopharyngeal carcinoma. Therefore, it is necessary to develop more-effective adjuvant therapies.

CIK cells (cytokine induced killer cells, CIK) are a population of heterogeneous cells generated by the in vitro amplification of mononuclear cells in peripheral blood. The cells are co-induced with multiple cytokines; the lymphocytes with co-expression of CD3+CD56+ have the strongest anti-tumor effect. Because of their non-MHC restricted tumor killing activity, CIK cells have a powerful anti-tumor effect both in vitro and in vivo, which spans a broad anti-tumor spectrum.

In this study, the patients with post-radiotherapy distant metastasis of NPC will be treated with autologous CIK cells in combination with Gemcitabine plus Cisplatin regimen chemotherapy(GC). The purpose of this study is to observe and evaluate the toxic side effects and the short- and long-term efficacy of CIK used in combination with GC chemotherapy to treat NPC in patients with distant metastasis after radiotherapy. Patients and Methods: 40 patients with distant metastasis after radiotherapy will accept 4 cycles chemotherapy of Gemcitabine plus cisplatin regimen and then are randomized divided into 2 groups. The 20 patients in GC+CIK group will be treated with maintaining therapy of adoptive autologous CIK cell transfusion sequentially; the other 20 patients will be followed-up only without CIK cells treatment. The safety of chemotherapy and CIK cells transfusion and the tumor regression status will be observed. The early response and long-term efficacy of two groups patients who accept GC chemotherapy or GC +CIK bio-therapy will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. The primary lesions of all patients were classified as undifferentiated, non-keratinizing carcinoma at the initial stage for treatment (WHO, 1991 criteria) and no distant metastasis was observed based on imaging studies before radiotherapy ;
2. all patients had received standard doses of radiotherapy, were regularly followed-up after radiotherapy, and had distant metastatic lesions revealed by imaging studies;
3. metastases were found more than 6 months after the end of radiotherapy, with the expected survival time of more than 3 months;
4. in each case, no more than 10 metastatic lesions were found in the imaging studies;
5. Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1;
6. the bone marrow functioned normally (WBC > 4.0×109/L, Hb > 120 g/L, PLT > 100×109/L);
7. the ECG results were normal, and the liver and kidney were functional.

Exclusion Criteria:

1. Patients were excluded if they had central nervous system metastases;
2. uncontrolled infection; underlying disease that was severe or life-threatening;
3. the patients were pregnant or lactating;
4. ECOG perform status ≥ 2;
5. the patients who are suffering from auto immune diseases or patients who need to accept glucocorticoid treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) | Participants will accept 4cycles GC regimen chemotherapy (every 4 weeks) plus 8 cycles CIK cells treatment (every 4 weeks), a total of therapy time will be 12 months.
  (According to the response criteria in solid tumor(RECIST), version 1.1)
  Complete remission (CR):Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial remission (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters;
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study ;
  Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Partial remission (PR) | Participants will accept 4cycles GC regimen chemotherapy (every 4 weeks) plus 8 cycles CIK cells treatment (every 4 weeks), a total of therapy time will be 12 months.
  (According to the response criteria in solid tumor(RECIST), version 1.1)
  Complete remission (CR):Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial remission (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters;
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study ;
  Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Stable disease (SD) | Participants will accept 4cycles GC regimen chemotherapy (every 4 weeks) plus 8 cycles CIK cells treatment (every 4 weeks), a total of therapy time will be 12 months.
  (According to the response criteria in solid tumor(RECIST), version 1.1)
  Complete remission (CR):Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial remission (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters;
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study ;
  Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Progressive disease (PD) | Participants will accept 4cycles GC regimen chemotherapy (every 4 weeks) plus 8 cycles CIK cells treatment (every 4 weeks), a total of therapy time will be 12 months.
  (According to the response criteria in solid tumor(RECIST), version 1.1)
  Complete remission (CR):Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial remission (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters;
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study ;
  Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).

SECONDARY OUTCOMES:
overall survival time (OS) | Paticipants will be follow-up 2 years afer they have accomplished 4 cycles GC chemotharapy /or GC chemotharapy plus CIK cells treatment.
  OS is defined as the time from randomization until death from any cause;
  TTP is defined as the time from randomization until objective tumor progression; TTP does not include deaths;
  PFS is defined as the time from randomization until objective tumor progression or death.
time to progression (TTP) | Paticipants will be follow-up 2 years afer they have accomplished 4 cycles GC chemotharapy /or GC chemotharapy plus CIK cells treatment.
  OS is defined as the time from randomization until death from any cause;
  TTP is defined as the time from randomization until objective tumor progression; TTP does not include deaths;
  PFS is defined as the time from randomization until objective tumor progression or death.
progression free survival(PFS) | Paticipants will be follow-up 2 years afer they have accomplished 4 cycles GC chemotharapy /or GC chemotharapy plus CIK cells treatment.
  OS is defined as the time from randomization until death from any cause;
  TTP is defined as the time from randomization until objective tumor progression; TTP does not include deaths;
  PFS is defined as the time from randomization until objective tumor progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China